CLINICAL TRIAL: NCT05485675
Title: Stand & Move at Work II: Effectiveness and Implementation of a Worksite Wellness Program
Acronym: SMWII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Minnesota (Other); The University of Queensland (Other); University of Nebraska (Other); University of Utah (Other); University of Virginia (Other)
Responsible Party: Principal Investigator, Matthew P Buman, PhD, Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01CA250527 (NIH); 1R01CA250527-01A1 (NIH)
Record Dates: First submitted 2021-12-01; First posted 2022-08-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Sedentary Behavior
Keywords: worksite health; sit-stand workstations; multilevel intervention; implementation science; fidelity; facilitation; effectiveness; sedentary behavior; posture; Light physical activity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: SMW and SMW+ will be running simultaneously.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stand & Move at Work (Active Comparator): Given an evidence-based workplace program to reduce sedentary behavior and increase standing and moving using a web-based platform. The web platform has a toolkit with strategies and guides for the worksite Champions to address changes at the environmental, social, and cultural levels.
  Interventions: Behavioral: Stand & Move at Work
- Stand & Move at Work+ (Experimental): This arm will receive access to the same web-based platform and toolkit as the other arm. Additionally, worksites in this arm will be assigned and expert facilitator who will meet regularly with the worksite Champions to assist with implementation.
  Interventions: Behavioral: Stand & Move at Work+

INTERVENTIONS:
Behavioral: Stand & Move at Work — Web-based platform only.
  Other Names: SMW
  Arms: Stand & Move at Work
Behavioral: Stand & Move at Work+ — Web-based platform and support from an expert facilitator
  Other Names: SMW+
  Arms: Stand & Move at Work+

SUMMARY:
This is a 2-arm group-randomized hybrid effectiveness-implementation (HEI type 2) study to test an evidence-based intervention (EBI) known as Stand & Move at Work(SMW) to reduce sedentary time in the workplace, and to test the role of expert facilitation (SMW+) for improving intervention fidelity.

DETAILED DESCRIPTION:
Primary Aim: To assess worksite-level reduction in sedentary time and intervention fidelity over 12 months Secondary Aim: To assess cost effectiveness of the intervention at 12 and 24 months

ELIGIBILITY:
Worksite-Level Inclusion Criteria:

* More than 80% of employees work full time (30+ hours per week).
* At least 45 employees in the worksite with sit-stand workstations working at least three days per week
* Occupations require primarily desk-based work (e.g., computer- and telephone-based)
* Willing to allow the researchers to distribute online research surveys to all employees in order to allow the program to be evaluated.
* Allow 30 randomly selected individuals to wear an activity monitor in several 7-day intervals across two years.
* Willing to be randomized to either intervention.
* Willing to identify one or more worksite champions to implement the Stand & Move at Work™ program.

Worksite-level exclusion criteria:

* Involved in previous interventions to reduce sitting and increase standing and moving at work in the last 24 months.
* Involved in the Stand and Move I intervention.
* Another worksite within the same organization is participating in the program and contamination across those worksites cannot be avoided.

Employee-level inclusion criteria:

* 18 years or older
* Willing to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4800 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Changes in posture | Baseline, 3 month, 12 months, and 24 months
  Accelerometer-based (activPAL) sensor fixed to the thigh that measures sitting, standing, and lying down over 7 days.
Competence/Adherence | 3 months
  A questionnaire-based assessment of intervention fidelity completed by study champions (competence and adherence) through an online portal. Based on Likert-scales and interval scales. SCORING RANGE
Competence/Adherence | 12 months
  A questionnaire-based assessment of intervention fidelity completed by study champions (competence and adherence) through an online portal. Based on Likert-scales and interval scales. SCORING RANGE
Competence/Adherence | 24 months
  A questionnaire-based assessment of intervention fidelity completed by study champions (competence and adherence) through an online portal. Based on Likert-scales and interval scales. SCORING RANGE
Intervention Fidelity | 3 months
  A questionnaire-based assessment of intervention fidelity completed by study participants regarding the advocates (competence and adherence) through an online portal. SCORING RANGE
Intervention Fidelity | 12 months
  A questionnaire-based assessment of intervention fidelity completed by study participants regarding the advocates (competence and adherence) through an online portal. SCORING RANGE
Intervention Fidelity | 24 months
  A questionnaire-based assessment of intervention fidelity completed by study participants regarding the advocates (competence and adherence) through an online portal. SCORING RANGE
Researcher derived measures of fidelity | 3 months
  A single composite measure of directly-observed intervention delivery assessed via web analytics, participation rates, and other calculated measures of fidelity.
Researcher derived measures of fidelity | 12 months
  A single composite measure of directly-observed intervention delivery assessed via web analytics, participation rates, and other calculated measures of fidelity.
Researcher derived measures of fidelity | 24 months
  A single composite measure of directly-observed intervention delivery assessed via web analytics, participation rates, and other calculated measures of fidelity.

SECONDARY OUTCOMES:
Comparison of program-related costs | Baseline, 3 month, 12 months, and 24 months.
  Program-related costs above and beyond cost of sit-stand workstation which may include advocate time spent implementing the intervention and intervention supplies.
Change in health-related quality of life | Baseline, 3 month, 12 months, and 24 months.
  36-Item Short Form Survey (SF36) assesses quality of life that will be used to estimate incremental cost effectiveness. Scored from 0 to 100, with 0 being maximum disability and 100 being no disability.
Change in musculoskeletal pain | Baseline, 3 months, 12 months, and 24 months.
  The Nordic Musculoskeletal Questionnaire (NMQ) assesses pain by bodily region on a Likert-type scale SCORING RANGE.
Change in Work Productivity and Activity Impairment Questionnaire - General Health | Baseline, 3 months, 12 months, and 24 months.
  Work Productivity and Activity Impairment Questionnaire: General Health (WPAI:GH) assesses impairment in paid work and activities in the preceding 7 days on an interval and Likert-type scale with a higher score indicating greater impariment.

OTHER OUTCOMES:
Change in sedentary behavior | Baseline, 3 month, 12 months, and 24 months.
  Sedentary behavior questionnaire (SBQ) is a brief questionnaire to assess time spent sitting in different work and non-work contexts SCORING RANGE

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Buman, PhD, Principal Investigator — Arizona State University College of Health Solutions; Mark Pereira, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Arizona State University College of Health Solutions, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Access to databases and associated software tools generated under the project will be available for educational, research and non-profit purposes. Such access will be provided using web-based applications, as appropriate. Publication of data shall occur during the project, if appropriate, and at the end of the project, consistent with normal scientific practices. Research data to document, support and validate research findings will be made available after the main findings from the final research data set have been accepted for publication. Such research data will be de-identified to prevent the disclosure of personal identifiers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Protocol and analysis plan will be available for sharing in 2022. Analytical code and data sets will be available for sharing following publication of the primary and secondary outcome papers.
Access Criteria: Public access via request to the study Principal Investigators